CLINICAL TRIAL: NCT01913561
Title: The Use of Master Caution Garment for Continuous Monitoring for Arrhythmia Detection Compared To Standard Gel-Electrode-Based ECG
Brief Title: The Use of Master Caution Garment for Continuous Monitoring for Arrhythmia Detection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HealthWatch Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HWG001
Record Dates: First submitted 2013-07-24; First posted 2013-08-01 (Estimated); Last update posted 2018-08-08 (Actual); Status verified 2018-08

CONDITIONS: Arrhythmia
Keywords: Electrocardiogram; gel electrodes; textile electrodes
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Master Caution Garment (Experimental): each patient will be connected simultaneously with two devices:
  * ECG gel electrodes
  * Master Caution Garment textile electrodes The two devices will be connected to hospital ECG telemetry.
  Interventions: Device: Master Caution Garment; Device: ECG gel electrodes

INTERVENTIONS:
Device: Master Caution Garment — Master Caution Garment is embedded with 10/13 textile dry electrodes that enable 12/15-lead ECG.
  The electrodes are dry, textile ECG electrodes.
  Other Names: MCG
Device: ECG gel electrodes — Standard gel electrodes that are been in use in hospital for ECG monitoring.

SUMMARY:
The Master Caution Garment is embedded with 10/13 textile dry electrodes that enable 12/15-lead ECG.

The electrodes are dry, textile ECG electrodes. The garment is designed to position the electrodes in the appropriate anatomical locations, without any special guidance. The dry electrodes are made from unique yarns with silver embedded into the garment using a proprietary technique developed by HealthWatch (HW)that obviates the need for skin preparation or the application of fluids. The garment can be connected to any standard ECG device available in the hospitals.

The purpose of this study is to evaluate the safety and effectiveness of the Master Caution Garment for continuous monitoring of ECG signal compared to standard gel electrodes.

The following endpoints will be evaluated in subjects participating in the study:

Primary:

Compare the quality of the ECG signal of HW textile electrodes compared to gel electrodes using standard ECG devices.

Secondary:

Compare the quality of the ECG signal of HW textile electrodes compared to gel electrodes when event is detected by the ECG devices.

DETAILED DESCRIPTION:
Part A - ECG in Rest

1. In the beginning of the study, the following parameters will be measured and documented in the CRF: blood pressure, body temperature, respiratory rate and oxygen saturation in the blood.
2. The patient will be dressed with the Master Caution Garment and connected to a 12 lead ECG device. The procedure takes 5 minutes including data printing.
3. A twelve lead ECG with gel electrodes will be done and data printed. The procedure takes 5 minutes. The patient will stay connected to the monitor for the following hour.
4. After an hour the data from the gel electrodes will be printed again.
5. The patient will be dressed again with the Master Caution Garment and connected to a 12 lead ECG device. The procedure takes 5 minutes including data printing.
6. The following parameters will be compared between the gel ECG and the Garment ECG:

   * Heart Rate (HR)
   * P wave width and amplitude
   * QRS complex width and amplitude
   * T wave width and amplitude
   * RR interval
   * PR interval
   * QT interval

Part B - ECG in motion

1. In the beginning of the study, the following parameters will be measured : blood pressure, body temperature, respiratory rate and oxygen saturation in the blood.
2. Four (4) gel electrodes will be placed on the patient on the following places - Left Arm (LA), Right Arm (RA), Left Leg (LL) and Right Leg (RL).
3. The patient will be dressed with the Master Caution Garment (MCG)on the 4 gel electrodes that were already placed.
4. The same 4 electrodes in the garment LA, RA, LL and RL will be connected to a standard of care ECG device.
5. The 4 gel electrodes will be connected to a standard of care ECG device.
6. The ECG devices will be recording the ECG signal from the two sets of electrodes for 24 hours.

   Every hour in the first 6 hours the data will be printed from both devices. In every event detected the data will be printed from both devices. the data will be evaluated for quality comparison between the gel and the textile electrodes using the hospital ECG device.
7. In first 6 hours for every hour and for each event detected by either the gel electrodes or the MCG textile electrodes the following parameters shell be evaluated at the end of the study from the hospital ECG printouts for the Master Caution Garment and for the gel electrodes:

   * Heart Rate (HR)
   * P wave width and amplitude
   * QRS complex width and amplitude
   * T wave width and amplitude
   * RR interval
   * PR interval
   * QT interval After first 6 hours for each event detected by either the gel electrodes or the MCG textile electrodes the above mentioned parameters shell be evaluated at the end of the study from the hospital ECG printouts for the Master Caution Garment and for the gel electrodes.

The goal of the current study is to evaluate the safety of the MCG and compare ECG signals from the Master Caution Garment with the ECG signals from gel electrodes.

This is a prospective, comparative study.

For each time interval and each event detected by the ECG devices, the analysis will determine its category as follows:

1. Blinded cardiologist's assessment whether at that time interval the patient suffered from a disorder. This assessment will be based on hospital's recorded data with the gel electrodes.
2. The Master Caution Garment result for that time interval will be categorized as follows:

   * True Positive (TP) = MCG Alert was right (based on GS)
   * False Positive (FP) = MCG Alert was wrong
   * True Negative (TN) = No MCG Alert when indeed alert was not necessary
   * False Negative (FN) = No MCG Alert but there was a disorder case

ELIGIBILITY:
Inclusion Criteria:

* Age>18 years.
* Suspected for arrhythmia or have evidence of arrhythmia disorder.
* Needs continuous, in-hospital ECG monitoring.
* Ability to give informed consent.

Exclusion Criteria:

* Patients with known allergy to silver.
* Patients with recent trauma to chest wall.
* Pregnant or lactating woman.
* Patients with chest deformity precluding placement of the garment.
* Patients participating in another ongoing trial.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2013-09; Primary Completion 2017-06 (Actual); Study Completion 2017-08-31 (Actual)

PRIMARY OUTCOMES:
From the ECG record collect the Heart Rate HR. | 0,1,2,3,4,5,6 hours and in each arrythemia event detected durring 24 hours from the start of the ECG recording.
From the ECG record collect the P Wave width (sec.) and the amplitude (mV). | 0,1,2,3,4,5,6 hours and in each arrythemia event detected durring 24 hours from the start of the ECG recording.
From the ECG record collect the QRS Complex width (sec.) and the amplitude (mV). | 0,1,2,3,4,5,6 hours and in each arrythemia event detected durring 24 hours from the start of the ECG recording.
From the ECG record collect the T Wave width (sec.) and the amplitude (mV). | 0,1,2,3,4,5,6 hours and in each arrythemia event detected durring 24 hours from the start of the ECG recording.
From the ECG record collect the RR Interval width (sec.). | 0,1,2,3,4,5,6 hours and in each arrythemia event detected durring 24 hours from the start of the ECG recording.
From the ECG record collect the PR Interval width (sec.). | 0,1,2,3,4,5,6 hours and in each arrythemia event detected durring 24 hours from the start of the ECG recording.
From the ECG record collect the QT Interval width (sec.). | 0,1,2,3,4,5,6 hours and in each arrythemia event detected durring 24 hours from the start of the ECG recording.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Zukerman, Dr., Principal Investigator — Rambam medical center Haifa, Israel
Locations (1):
- Rambam medical center, Haifa, Israel